CLINICAL TRIAL: NCT07375004
Title: Adjunctive Use of Injectable PRF in Non-surgical Periodontal Therapy: Clinical and Microbiological Outcomes ( Split - Mouth Randomized Controlled Trial )
Brief Title: Injectable PRF in Non-Surgical Periodontal Treatment
Acronym: IPRF-PERIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Thuraya ayad taher al-jubori, Master student, Al-Mustansiriyah University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UOM-DENT-ETHIC-2026-042
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Periodontal Pocket; Alveolar Bone Loss
Keywords: Injectable Platelet-Rich Fibrin; i-PRF; Scaling and Root Planing; Non-Surgical Periodontal Therapy; Split-mouth design; Microbiological outcomes; Periodontitis; Regeneration
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Alveolar Bone Loss | interventions — proliferation regulatory factors, human urine; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: This is a split-mouth randomized controlled trial. Each participant receives both treatments in different quadrants of the mouth. One quadrant is randomly assigned to the intervention (Scaling and Root Planing + i-PRF) and the contralateral quadrant serves as the control (Scaling and Root Planing alone)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study follows a double-blind protocol regarding outcome assessment and data analysis. The clinical and microbiological examiner (Outcomes Assessor) is masked to the treatment allocation. Furthermore, the statistician (Statistical Investigator) will receive the data in a coded format (e.g., Side A and Side B) without knowing which side received the i-PRF intervention until the final analysis is completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: i-PRF + SRP (Experimental): This quadrant of the mouth will receive full-mouth scaling and root planing (SRP) followed by the subgingival injection of injectable Platelet-Rich Fibrin (i-PRF) into the periodontal pockets
  Interventions: Biological: Injectable Platelet-Rich Fibrin (i-PRF).; Procedure: Scaling and Root Planing (SRP).
- Active Comparator: SRP Alone (Active Comparator): This contralateral quadrant of the mouth will receive full-mouth scaling and root planing (SRP) only, serving as the control side to compare with the i-PRF intervention.
  Interventions: Procedure: Scaling and Root Planing (SRP).

INTERVENTIONS:
Biological: Injectable Platelet-Rich Fibrin (i-PRF). — Ten ml of whole blood is collected from the participant into plain tubes and immediately centrifuged. The centrifugation protocol follows the low-speed concept (e.g., 700 rpm for 3 minutes). The upper orange-colored liquid (i-PRF) is then collected and injected subgingivally into the periodontal pockets using a 25-gauge needle immediately after scaling and root planing
  Other Names: Autologous Platelet Concentrate.; i-PRF
  Arms: Experimental: i-PRF + SRP
Procedure: Scaling and Root Planing (SRP). — Full-mouth non-surgical periodontal therapy including supra and sub-gingival scaling and root planing performed using ultrasonic devices and Gracey curettes to remove dental biofilm and calculus
  Other Names: Non surgical periodontal therapy; SRP; Initial periodontal therapy; Phase I periodontal therapy; Cause related periodontal therapy

SUMMARY:
This study aims to evaluate the clinical and microbiological effects of using injectable Platelet-Rich Fibrin (i-PRF) as an adjunct to non-surgical periodontal therapy (scaling and root planing) in patients with periodontitis. The study uses a split-mouth design where one side of the mouth receives the treatment with i-PRF and the other side receives standard treatment alone. Clinical parameters and bacterial counts will be compared at baseline, 1 month, and 3 months after intervention .

DETAILED DESCRIPTION:
Patients with periodontitis will be recruited for this split-mouth randomized controlled trial. All participants will receive full-mouth supra and sub-gingival scaling and root planing (SRP). In the intervention side, i-PRF will be injected into the periodontal pockets, while the control side will receive SRP only.

Clinical measurements including Probing Pocket Depth (PPD), Clinical Attachment Level (CAL), and Bleeding on Probing (BOP) will be recorded. Additionally, microbiological samples will be collected to assess the changes in the subgingival Porphyromonas gingivalis and Fusobacterium nucleatum . Follow-up visits are scheduled at 1 and 3 months post-intervention to assess the adjunctive benefit of i-PRF.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 30 years and above.
* No history of systemic diseases (e.g., diabetes mellitus).
* Not currently under active periodontal therapy or joining other trial in the last 3 months.
* Diagnosis with Stage II or III Periodontitis.
* presence of interdental CAL affecting ≥2 non adjacent teeth or if CAL at buccal/lingual aspects associated with PPD >4mm at ≥2 teeth.

Exclusion Criteria:

* Smokers or alcohol users.
* Patients consuming antibiotics or anticoagulants.
* Regular users of non-steroidal anti-inflammatory drugs.
* Receipt of periodontal treatment within 3 months prior to the study.
* Any bleeding or clotting disorders.
* Teeth with Grade II or Grade III furcation involvement.
* Pregnant or breastfeeding mothers.
* Patients unwilling to participate.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline, 1 month, and 3 months post-intervention
  Probing pocket depth will be measured in millimeters from the gingival margin to the base of the periodontal pocket using a standardized periodontal probe (e.g., William's probe) at six sites per tooth.

SECONDARY OUTCOMES:
Clinical Attachment Level (CAL) | Baseline, 1 month, and 3 months post-intervention
  Measurement of the distance from the cemento-enamel junction (CEJ) to the base of the periodontal pocket in millimeters.
Bleeding on Probing (BOP) | Baseline, 1 month, and 3 months post intervention
  Assessment of the presence or absence of bleeding within 30 seconds after probing, recorded as a percentage of total sites.
Plaque Index (PI) | Baseline, 1 month, and 3 months post intervention .
  Assessment of the amount of dental plaque on the tooth surfaces to evaluate the patient's oral hygiene during the study.
Microbiological Analysis (Bacterial Load) | Baseline, 1 month, and 3 months post intervention
  Quantification of subgingival periodontal pathogens (P. gingivalis and F. nucleatum )using Quantitative Real-time PCR (qPCR) from subgingival plaque samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustansiriyah University, College of Dentistry., Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No